CLINICAL TRIAL: NCT06911892
Title: Cutaneous Sensory Mapping and Comparative Analysis of Different Regional Anesthesia Techniques in Breast Cancer Surgeries: A Prospective Observational Study
Brief Title: Comparative Sensory Mapping of Regional Anesthesia Techniques in Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2025/6/11
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Pain, Postoperative
Keywords: Regional Anesthesia; Pain Management; Cutaneous Sensory Mapping
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group Serratus Anterior Plane Block: Patients who received ultrasound-guided Serratus Anterior Plane Block during the preoperative period.
  Interventions: Other: Group Serratus Anterior Plane Block
- Group Parasternal Block: Patients who received ultrasound-guided Parasternal Block during the preoperative period.
  Interventions: Other: Group Parasternal Block
- Group Interpectoral+Pectoserratus Plane Block: Patients who received ultrasound-guided Interpectoral+Pectoserratus Plane Block during the preoperative period.
  Interventions: Other: Group Interpectoral+Pectoserratus Plane Block

INTERVENTIONS:
Other: Group Serratus Anterior Plane Block — Patients will receive a serratus anterior plane block preoperatively under ultrasound guidance. Thirty minutes after the block, the cutaneous sensory area will be assessed using a pinprick test and outlined on the skin using a UV marker. Subsequently, the incision line for the modified radical mastectomy (MRM) will be marked by the operating surgeon. The resulting drawings will be documented and transferred to a digital template for analysis.
  Groups: Group Serratus Anterior Plane Block
Other: Group Parasternal Block — Patients will receive a parasternal block preoperatively under ultrasound guidance. Thirty minutes after the block, the cutaneous sensory area will be assessed using a pinprick test and outlined on the skin using a UV marker. Subsequently, the incision line for the modified radical mastectomy (MRM) will be marked by the operating surgeon. The resulting drawings will be documented and transferred to a digital template for analysis.
  Groups: Group Parasternal Block
Other: Group Interpectoral+Pectoserratus Plane Block — Patients will receive an interpectoral + pectoserratus plane block preoperatively under ultrasound guidance.
  Thirty minutes after the block, the cutaneous sensory area will be assessed using a pinprick test and outlined on the skin using a UV marker. Subsequently, the incision line for the modified radical mastectomy (MRM) will be marked by the operating surgeon. The resulting drawings will be documented and transferred to a digital template for analysis.
  Groups: Group Interpectoral+Pectoserratus Plane Block

SUMMARY:
Various regional anesthesia techniques, either individually or in combination, can be utilized for analgesia in breast cancer surgery. This study aims to map the cutaneous sensory block areas of different regional anesthesia techniques (serratus anterior plane block, parasternal block, and interpectoral + pectoserratus plane block) applied to patients undergoing breast cancer surgery. Furthermore, the extent to which these blocks cover the modified radical mastectomy incision will be assessed. The study seeks to comparatively determine the minimum and maximum sensory spread of each block. Ultimately, the findings are intended to provide valuable data for developing tailored perioperative pain management strategies specific to the surgical procedure and individual patient needs.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women, and surgical intervention is frequently employed as a treatment modality. However, the choice of surgical approach may vary depending on the tumor subtype and the extent of metastasis. The orientation of the surgical incision also differs based on the tumor location and/or the presence of axillary involvement.

Accurately identifying the anatomical location of the affected tissues during breast surgery is of critical importance for planning an effective perioperative analgesia strategy. Procedures such as lumpectomy, partial mastectomy, and therapeutic mammoplasty primarily involve the skin and subcutaneous breast tissue. Depending on whether the surgery is performed medial or lateral to the nipple, the anterior or lateral cutaneous branches of the intercostal nerves play a role in innervating the surgical area. In more extensive surgeries such as modified radical mastectomy (MRM), nerves originating from the brachial plexus (pectoralis, thoracodorsal, and long thoracic nerves) may contribute to perioperative pain. These procedures typically involve the dissection of all subcutaneous breast tissue, the overlying skin, and the pectoralis and serratus anterior muscles and often necessitate sentinel lymph node biopsy or axillary dissection.

Due to these factors, various incision types are used in oncological breast surgeries depending on the type of surgery. Therefore, a patient-specific perioperative pain protocol should be established for each procedure, and the most appropriate regional anesthesia technique should be selected accordingly.

In the literature, serratus plane blocks, paravertebral block, interpectoral, and pectoserratus blocks, as well as their combination, have been reported to provide effective perioperative pain management in breast cancer surgery. These techniques offer benefits such as reducing acute and chronic pain, minimizing the surgical stress response, facilitating early mobilization, decreasing opioid consumption, and ensuring a more hemodynamically stable perioperative period.

In the investigators' clinic, regional anesthesia techniques guided by ultrasound are routinely administered, either alone or in combination, to manage perioperative pain in patients undergoing breast cancer surgery. These techniques include serratus anterior plane block, parasternal block, and interpectoral + pectoserratus plane block.

The study was designed as an observational clinical trial to evaluate patients undergoing breast cancer surgery who received regional anesthesia for perioperative pain management. The primary objective is to evaluate the cutaneous sensory block areas of these blocks and compare the blocked sensory areas with the modified radical mastectomy incision to assess the minimum and maximum sensory spread of each block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral breast cancer surgery
* Patients receiving regional anesthesia as part of their perioperative analgesia management
* Aged between 18 and 70 years.
* ASA<IV
* Patients who agree to participate and provide written informed consent

Exclusion Criteria:

* Patients who refuse to participate.
* Patients who have not undergone any regional anesthesia technique.
* ASA>III
* Bilateral mastectomy.
* History of previous breast surgery (except excisional biopsy).
* Cognitive impairment or dementia.
* Patients with psychiatric disorders such as depression, mania, or schizophrenia.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients scheduled for breast cancer surgery will be included.
Study Population: Patients scheduled for breast cancer surgery and receiving regional anesthesia as part of their perioperative analgesia management will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Cutaneous sensory block area mapping for different regional anesthesia techniques in breast cancer surgery | At 30 minutes after the regional anesthesia and before surgery
  The cutaneous sensory block area resulting from the regional anesthesia technique applied to each patient will be assessed using a pinprick test at the 30th minute post-block. These areas will be delineated and mapped using a UV marker, and the data collected for each group will be processed to generate a density map using the digital template.

SECONDARY OUTCOMES:
Determination of the minimum and maximum spread of each block technique in relation to the modified radical mastectomy (MRM) incision | At 30 minutes after the regional anesthesia and before surgery
  The cutaneous sensory block area following the regional anesthesia technique will be compared with the modified radical mastectomy (MRM) incision indicated by the surgeon on the patient. The images will be documented and analyzed with digital template. Areas that correspond (either fully or partially) with the incision line will be identified. For each block technique, the minimum and maximum spread of the modified radical mastectomy (MRM) incision will be determined and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Caner Genc, M.D., Study Director — Samsun University
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] FitzGerald S, Odor PM, Barron A, Pawa A. Breast surgery and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):95-110. doi: 10.1016/j.bpa.2019.03.003. Epub 2019 Apr 6. PMID 31272657
- [Background] Hargrave J, Grant MC, Kolarczyk L, Kelava M, Williams T, Brodt J, Neelankavil JP. An Expert Review of Chest Wall Fascial Plane Blocks for Cardiac Surgery. J Cardiothorac Vasc Anesth. 2023 Feb;37(2):279-290. doi: 10.1053/j.jvca.2022.10.026. Epub 2022 Nov 1. PMID 36414532
- [Background] Jacobs A, Lemoine A, Joshi GP, Van de Velde M, Bonnet F; PROSPECT Working Group collaborators#. PROSPECT guideline for oncological breast surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2020 May;75(5):664-673. doi: 10.1111/anae.14964. Epub 2020 Jan 26. PMID 31984479